CLINICAL TRIAL: NCT01409733
Title: TACE With Drug Eluting Beads Loaded With Doxorubicin in Liver Metastases From Melanoma Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: University Hospital Tuebingen (Other); SLK Kliniken Heilbronn GmbH (Other)
Responsible Party: Prof. Philippe Pereira, SLK Klinikum Heilbronn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pereira-DE-2010
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: Stage IV Melanoma Patients With Unresectable Liver Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stage IV melanoma patients (Experimental)
  Interventions: Device: TACE using Drug Eluting Beads loaded with Doxorubicin

INTERVENTIONS:
Device: TACE using Drug Eluting Beads loaded with Doxorubicin — 100-300 microns DC Beads loaded with Doxorubicin (75mg of Doxorubixcin per vial)
  Other Names: DC Bead; DebDox

SUMMARY:
The Aim is to evaluate safety and efficacy of TACE with doxorubicin-loaded DC beads in melanoma patients with liver metastasis. This is a pilot study with the aim of recruiting 20 patients, this is a feasibility study. the patients profile is patients with stage IV Melanoma with liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable, measurable disease defined as at least one lesion that can be accurately and serially measured per the modified RECIST and EASL criteria (2D/3D-EASL) or MRI (Extent of Necrosis)
2. Patients ≥ 18 years of age, > 35kg, of any race or sex, who have histological or radiological proof of melanoma to the liver
3. ECOG performance status < 3.
4. Patient chooses to participate and has signed the informed consent document.
5. Patients with unilobar disease who can be treated superselectively in a single session or patients with bilobar disease who can have both lobes able to be treated within 3 - 4 weeks in separate sessions.
6. Patients with patent main portal vein.
7. Ocular melanoma is allowed.
8. Patients with clinically and radiologically stable brain metastasis from melanoma can be included.
9. Patients with liver dominant disease (>50% overall tumor burden).
10. Prior systemic therapy for metastatic disease is allowed.
11. Non-pregnant with an acceptable contraception in premenopausal women and fertile men.
12. Hematological function: ANC ≥1.5 x 109/L, platelets ≥ 75 x 109/L, INR<1.3 (patients on therapeutic anticoagulants are not eligible).
13. Adequate renal function: Creatinine ≤2.0mg/dl and GFR >30.
14. Adequate liver function: total bilirubin ≤ 2.5 mg/dl, ALT, AST ≤ 5 times ULN, albumin ≥ 2.5mg/dl.
15. All toxic effects of prior therapy must have resolved to ≤ Grade 1 unless otherwise specified above

Exclusion Criteria:

1. Women who are pregnant or breast feeding.
2. Patients eligible for curative treatment such as resection or radiofrequency ablation.
3. Active bacterial, viral or fungal infection within 72 hours of study entry.
4. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (TA, Tis & Ti) or any cancer curatively treated < 5 years prior to study entry.
5. Contraindication to hepatic artery embolization procedures:

   - Severe peripheral vascular disease precluding catheterization.
6. - Large shunt as determined by the investigator (pretesting with TcMAA not required) at the time of first angiogram.
7. -Hepatofugal blood flow.
8. -Main portal vein occlusion (e.g. thrombus or tumor).
9. Recovery from major trauma including surgery within 4 weeks prior to administration of study treatment.
10. Allergy to contrast media that cannot be managed with standard care (e.g. steroids), making magnetic resonance imaging (MRI) or computed tomography (CT) contraindicated.
11. Advanced liver disease (> 80% liver replacement).
12. Other significant medical or surgical condition, or any medication or treatment that would place the patient at undue risk and that would preclude the safe use of chemoembolization or would interfere with study participation.
13. Ongoing systemic cancer treatment.
14. Any contraindication for Doxorubicin administration:
15. WBC <3000 cells/mm3
16. Neutrophils <1500 cells/mm3
17. Deficient cardiac function defined as a LVEF of <50% normal
18. Allergy to Doxorubicin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients completing scheduled treatment plan | 12 months
  Safety: Adverse Events Efficacy: Response to Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Pereira, MD, Principal Investigator — SLK Klninikum
Locations (1):
- SLK Klinikum, Heilbronn, Germany